CLINICAL TRIAL: NCT00144014
Title: A Phase II, Multi-centre, Two-part Study to Evaluate the Safety and Efficacy of Study Drug in Acute Ischaemic Stroke.
Brief Title: Safety and Efficacy Study in Acute Ischaemic Stroke
Acronym: VASST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V10153-2S-01
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Stroke
Keywords: Acute; Ischaemic; Stroke
MeSH Terms: conditions — Stroke; Ischemia | interventions — BB-10153

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- V10153, 1.0 mg/kg (Experimental): Single acute intravenous bolus dose
  Interventions: Drug: V10153
- V10153, 2.5 mg/kg (Experimental): Single acute intravenous bolus dose
  Interventions: Drug: V10153
- V10153, 5.0 mg/kg (Experimental): Single acute intravenous bolus dose
  Interventions: Drug: V10153
- V10153, 7.5 mg/kg (Experimental): Single acute intravenous bolus dose
  Interventions: Drug: V10153
- V10153, 10 mg/kg (Experimental): Single acute intravenous bolus dose
  Interventions: Drug: V10153

INTERVENTIONS:
Drug: V10153 — Single acute intravenous bolus dose up to 10 mg/kg
  Other Names: Code Names: V10153, BB-10153; CAS Registry Number: 931101-84-7; Proposed INN: Troplasminogen alfa

SUMMARY:
A Phase II study to evaluate the safety and efficacy of five dose levels of study drug in acute ischaemic stroke

DETAILED DESCRIPTION:
An open label, dose escalation study where patients with acute ischaemic stroke will receive a single intravenous dose of study drug. There will be five dose levels with groups of 10 patients in each. Escalation to higher doses will occur following review of safety data from the previous dose.

ELIGIBILITY:
Summary of Inclusion Criteria:

1. Onset of new neurological signs of stroke within 3 to 9 hours of the time to initiation of treatment
2. Aged 18 and above
3. Provide consent
4. Cerebral CT scan to show findings of early ischaemic changes consistent with the clinical diagnosis and an ASPECT score of between 5 and 10 inclusive.
5. NIHSS score greater than 5 or less than or equal to 20.

Summary of Exclusion Criteria:

1. Coma
2. Stroke with unknown time of onset
3. Minor stroke symptoms and sings (<6 points on the NIHSS) which are rapidly improving by the time of randomisation.
4. Major stroke symptoms and signs (>20 on the NIHSS)
5. History of stroke in previous 6 weeks
6. History of brain tumours
7. CT scan results in an ASPECT score of <5
8. Haemorrhagic risk
9. Abnormal laboratory values
10. Positive urine pregnancy test, lactation or parturition within previous 30 days.
11. Weight >135 kg
12. Uncontrolled hypertension.
13. Raised blood glucose
14. History of or current serious illness
15. Participation in another clinical trial within 4 weeks of drug administration

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-08; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To establish the safety of five dose levels (1.0, 2.5, 5, 7.5 and 10 mg/kg)of V10153 in patients with acute ischaemic stroke. | Ongoing

SECONDARY OUTCOMES:
To compare recanalisation rates across dose levels. | Ongoing
To compare clinical outcome between treatments by NIHSS, Modified Rankin Scale and Barthel Index. | Post-study completion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hill, Principal Investigator — Foothills Hosptial
Locations (28):
- United States (23):
  - Stroke Centre, Mayo Clinic, Scottsdale, Arizona
  - UCLA Stroke Network, Los Angeles, California
  - Neurology Medical Group of Diablo Valley, Walnut Creek, California
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Bradenton Research Centre, Bradenton, Florida
  - Ocala Neurodiagnostic Centre, Ocala, Florida
  - Florida Hospital of Neuroscience Institute, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Florida Neurovascular Institue Stroke Center, Tampa, Florida
  - Vascular Neurology, Loyola University Medical Center, Maywood, Illinois
  - Center for Advanced Medicine, Jewish Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - UMAS Memorial Medical Centre, Worcester, Massachusetts
  - Sunrise Hospital and Medical Centre, Las Vegas, Nevada
  - Washoe Stroke Center, Reno, Nevada
  - Stroke Centre, Neurological Institute, Carolinas Medical Centre, Charlotte, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Medical University South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - Neurological Institute, The Methodist Hospital, Houston, Texas
  - Division of Neuro-Ophthalmology, Virginia Commonwealth University, Richmond, Virginia
- Canada (5):
  - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Centre for Stroke Research, Vancouver Island Health Research Centre, Victoria, British Columbia
  - 71 King Street West, Mississauga, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Hospital Charles LeMoyne, Québec

IPD SHARING:
Plan to Share IPD: Undecided